CLINICAL TRIAL: NCT02618265
Title: Mobile Terminal Based Management and Platelet Reactivity Modified Drug Regulation of Stroke Secondary Prevention
Brief Title: Mobile Terminal Based Management of Stroke Secondary Prevention Adminstration Effect Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Fan Dongsheng, Chairman of Neurology Department, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUTH2013144
Record Dates: First submitted 2015-09-16; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: stroke; secondary prevention; platelet response polymorphism; mobile terminal
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobile terminal (Experimental): Stroke received mobile terminal management for secondary prevention administration, as the same time platelet reactivity modified drug selection was performed. Mobile application management conducts the control and regulation for anti hypertension, statin and antiplatelet therapy to increasing drug compliance.
  Interventions: Procedure: Mobile terminal
- traditional management (Active Comparator): Stroke received traditional management for secondary prevention administration
  Interventions: Procedure: traditional management
- website platform management (Active Comparator): Stroke received website platform management for secondary prevention administration. Website platform management conducts the control and regulation for anti hypertension, statin and antiplatelet therapy to increasing drug compliance.
  Interventions: Procedure: website platform management

INTERVENTIONS:
Procedure: Mobile terminal — multiple strategy including mobile terminal based compliance managment, platelet reactivity modified drug adjustment
  Other Names: Mobile Application
  Arms: Mobile terminal
Procedure: traditional management — aspirin or clopidogrel monotherapy or double treatment for
  Other Names: traditional second prevention
  Arms: traditional management
Procedure: website platform management — second prevention based on website platform management
  Arms: website platform management

SUMMARY:
The investigators want to verify whether mobile application based on stroke strengthen prevention management is more effective than traditional management model or open stroke management platform. Whole blood-impedance based platelet aggregation(WBA) method and VerifyNow detected by aspirin or clopidogrel responsiveness will provide individualized anti-platelet drug selection. Endpoint event is defined as stroke death or relapse. Primary measure outcomes are change of the stroke recurrence rate and mortality after secondary prevention.

DETAILED DESCRIPTION:
With high incidence, mortality, morbidity and recurrence rate，stroke has significant impact on national development strategies planning. Improving secondary prevention will strongly promote stroke management in the rapid developing phase of Chinese economy and expansion of health situation. At present lack of high-quality medical resources, low medical permeability cannot remedy extensive prevention failure of stroke. Mobile healthcare is easier to conduct and still in the early stage of explosive growth. This research group has established an open management platform of stroke prevention. And collaborate with Peking University Institute of Information Technology to develop a smart phone application which can be personalized medication reminder, record medication compliance, home blood pressure and blood glucose test results, also can provide doctor-patient communication platform and symptoms alarm. The investigators want to verify whether mobile application based on stroke strengthen prevention management is more effective than traditional management model or open stroke management platform. Whole blood-impedance based platelet aggregation(WBA) method and VerifyNow detected by aspirin or clopidogrel responsiveness will provide individualized anti-platelet drug selection. Control group will be selected from the National Stroke data registration database platform and open platform for stroke prevention. Follow-up period is 2 years. Endpoint event is defined as stroke death or relapse. Primary measure outcomes are change of the stroke recurrence rate and mortality after secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* stroke

Exclusion Criteria:

* refusion in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change of the stroke recurrence rate | 2 years stroke recurrence rate
  After secondary prevention

SECONDARY OUTCOMES:
change of the stroke mortality | 2 years stroke mortality
  After secondary prevention

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Study Director — PUTH
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Y, Fan D, Qiao S, Hu H. Verifynow P2Y12 PRU-Guided Modification of Clopidogrel for Prevention of Recurrent Ischemic Stroke: A Real-World Prospective Cohort Study. Neurol Ther. 2022 Dec;11(4):1749-1766. doi: 10.1007/s40120-022-00406-z. Epub 2022 Sep 26. PMID 36163415
- [Derived] Zhang Y, Fan D, Ji H, Qiao S, Li X. Treatment Adherence and Secondary Prevention of Ischemic Stroke Among Discharged Patients Using Mobile Phone- and WeChat-Based Improvement Services: Cohort Study. JMIR Mhealth Uhealth. 2020 Apr 15;8(4):e16496. doi: 10.2196/16496. PMID 32293574